CLINICAL TRIAL: NCT02720328
Title: Prevalence and Causes of Preventable and Serious Adverse Drug Reactions Related to the Use of Oral Anticoagulants
Acronym: ADR-OAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: v6
Record Dates: First submitted 2016-03-07; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Embolism and Thrombosis; Hemorrhage
MeSH Terms: conditions — Embolism and Thrombosis; Hemorrhage | interventions — Blood Specimen Collection

ARMS (1):
- DOAC-treated patients (Other): Concerning patients taking DOACs, blood samples are drawn to evaluate DOAC plasma concentration. One EDTA tube is also drawn to extract DNA and determine the genetic profile of genes involved in the metabolism of DOACs. The aim will be to assess if genetic determinants can explain the observed interindividual variability in plasma concentrations.
  Interventions: Biological: Blood samples for DOAC measurement

INTERVENTIONS:
Biological: Blood samples for DOAC measurement

SUMMARY:
The purpose of this study is to investigate the preventability of serious adverse drug reactions (ADRs) related to the use of direct oral anticoagulants (DOACs). The investigators also aim at identifying the underlying causes of these preventable ADRs. The endpoint measurements will be compared with a group of patients taking vitamin-K antagonists (VKAs). For this purpose, a protocol for a prospective observational study was developed. The study was approved by the Ethics Committee of the CHU UCL Namur (site Godinne) and the Cliniques Universitaires Saint-Luc. Patients admitted to the emergency department of these two teaching hospitals with a thrombotic or a bleeding event while under DOAC or VKA are included. After a comprehensive medication history, the appropriateness of prescribing is evaluated, using an adapted version of the Medication Appropriateness Index. Causality, severity and preventability of adverse events are assessed by two pharmacists and two hematologists using predefined scales. Second, for cases of serious and preventable ADRs, semi-structured interviews are performed with general practitioners to understand the underlying causes of medication errors. Based on the results, risk-minimization strategies that specifically target the problems encountered in clinical practice will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the emergency department
* Presenting a thrombotic or a bleeding event
* Prescribed NOAC (rivaroxaban, dabigatran etexilate or apixaban) or VKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Preventability of adverse drug reactions according to Hallas criteria | Baseline

SECONDARY OUTCOMES:
Appropriateness of prescribing according to the Medication Appropriateness Index | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU UCL Namur site Godinne, Yvoir